CLINICAL TRIAL: NCT03726372
Title: Effect of Neuromuscular Blockade Protocol on Perioperative Outcomes of Robotic Laparoscopic Surgery
Brief Title: Muscle Relax Affects Outcomes of Robotic Surgery
Acronym: MORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, principle investigator, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-20180701
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: General Anesthesia; Postoperative Complications
Keywords: robotic surgery; laparoscopic surgery; neuromuscular blockade; postoperative complication
MeSH Terms: conditions — Postoperative Complications | interventions — Rocuronium; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Muscle relaxant will be given by a specific investigator that is not involved in anesthesia and outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep neuromuscular blockade (Experimental): Rocuronium, a neuromuscular blocking agent will be given by continuous infusion at a dose that reaction to train of four (TOF) stimulation is depressed to zero
  Interventions: Drug: Rocuronium; Other: continuous infusion
- moderate neuromuscular blockade (Experimental): Rocuronium, a neuromuscular blocking agent will be given at a dose by intermittent injection that reaction to train of four (TOF) stimulation is kept 1 to 2
  Interventions: Drug: Rocuronium; Other: intermittent injection

INTERVENTIONS:
Drug: Rocuronium — rocuronium is a neuromuscular blocking agent with a duration of 40 minutes
  Other Names: rocuronium bromide
Other: continuous infusion — rocuronium is continuously infused
  Other Names: high dose
  Arms: deep neuromuscular blockade
Other: intermittent injection — rocuronium is intermittently given
  Other Names: low dose
  Arms: moderate neuromuscular blockade

SUMMARY:
During robotic laparoscopic surgery, a high intraperitoneal pressure may result in high airway pressure and inadequate perfusion of the abdominal organs, and as a result the postoperative outcomes. Degree of neuromuscular blockade (NMB) can affect the intraperitoneal pressure. In this study, the patients undergoing robotic laparoscopic surgery will be assigned to deep NMB group and moderate NMB group. Perioperative outcomes including maximal intraperitoneal pressure, maximal intraoptic pressure, quality of emergence, postoperative pain, and incidence of postoperative respiratory complication will be compared. The results of this study will provide evidence for optimizing NMB protocol of robotic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective robotic laparoscopic surgery under general anesthesia
* American Society of Anesthesiologists status 1-2
* Body mass index of 18-30kg/m2
* Patients scheduled to be positioned in trendelenburg position during surgery

Exclusion Criteria:

* Patients allergic to rocuronium
* Patients with neuromuscular dysfunction
* Patients with existed pulmonary diseases
* Patients with hepatic or renal dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-11-10 (Estimated); Study Completion 2019-11-10 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative major respiratory complications | from end of surgery to discharge, at an average of 4 days
  incidence of pneumonia and atelectasis

SECONDARY OUTCOMES:
maximal airway pressure | from establishment of pneumoperitoneum to end of pneumoperitoneum, at an average of 3 hours
  airway pressure is titrated to as low as possible as long as the end tidal carbon dioxide partial pressure is lower than 40 mmHg
minimal cerebral oxygen saturation | from start of surgery to end of surgery, at an average of 3.5 hours
  cerebral oxygen saturation is continuously monitored during surgery
maximal intraocular pressure | from start of surgery to end of surgery, at an average of 3.5 hours
  intraocular pressure is monitored every 10 minutes during surgery
number of surgeon asking for improving muscle relax | from start of surgery to end of surgery, at an average of 3.5 hours
  when the surgeon is unsatisfied with the muscle relax, he can tell the anesthetist
time to extubation | from end of sevoflurane inhalation to extubation, at an average of 20 minutes
  criteria of extubation: spontaneous respiratory rate>10 per minute and end tidal carbon dioxide partial pressure<45mmHg
incidence of nausea and vomiting in post-anesthesia care unit | from admittance to post-anesthesia care unit(PACU) to discharge from PACU, at an average of 30 minutes
incidence of shoulder pain in 24 hours after surgery | from end of surgery to 24 hours after surgery
incidence of residual neuromuscular blockade in the post-anesthesia care unit | from admittance to post-anesthesia care unit(PACU) to discharge from PACU, at an average of 30 minutes
  residual neuromuscular blockade is defined as time of head-lift or limb-lift<10 seconds
visual analogue scale at 24 hours after surgery | end of surgery to 24 hours after surgery
  the patients are asked to mark the score they feel, 0 is no pain,100 is untolerated pain
expense after surgery | end of the surgery to discharge,at an average of 4 days
  the expense from immediately after surgery to discharge
satisfaction score of the patients | from end of surgery to discharge,at an average of 4 days
  the patient is asked to give a score between 0 and 10, 0 means not satisfied,10 means totally satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Lu, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Yes
After publishing, data of the primary endpoint and second endpoints can be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When the results have been published in peer-reviewed journals, the data will be available. The planned time frame will be 5 years.

REFERENCES:
- [Background] Van Wijk RM, Watts RW, Ledowski T, Trochsler M, Moran JL, Arenas GW. Deep neuromuscular block reduces intra-abdominal pressure requirements during laparoscopic cholecystectomy: a prospective observational study. Acta Anaesthesiol Scand. 2015 Apr;59(4):434-40. doi: 10.1111/aas.12491. Epub 2015 Feb 13. PMID 25684372
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Barrio J, Errando CL, Garcia-Ramon J, Selles R, San Miguel G, Gallego J. Influence of depth of neuromuscular blockade on surgical conditions during low-pressure pneumoperitoneum laparoscopic cholecystectomy: A randomized blinded study. J Clin Anesth. 2017 Nov;42:26-30. doi: 10.1016/j.jclinane.2017.08.005. Epub 2017 Aug 30. PMID 28803124
- [Background] Torensma B, Martini CH, Boon M, Olofsen E, In 't Veld B, Liem RS, Knook MT, Swank DJ, Dahan A. Deep Neuromuscular Block Improves Surgical Conditions during Bariatric Surgery and Reduces Postoperative Pain: A Randomized Double Blind Controlled Trial. PLoS One. 2016 Dec 9;11(12):e0167907. doi: 10.1371/journal.pone.0167907. eCollection 2016. PMID 27936214